CLINICAL TRIAL: NCT00756821
Title: A Pilot Study of Biomarkers for Spinal Muscular Atrophy
Acronym: BforSMA
Status: Completed | Type: Observational
Sponsor: Carelon Research (Other)
Collaborators: The Spinal Muscular Atrophy Foundation (Other)
Responsible Party: The Spinal Muscular Atrophy Foundation, The Spinal Muscular Atrophy Foundation
Other Study IDs: BforSMA
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy; Blood Biomarkers; Urine Biomarkers; Type I Spinal Muscular Atrophy; Type II Spinal Muscular Atrophy; Type III Spinal Muscular Atrophy; Modified Hammersmith Functional Motor Scale; Disease severity; Biomarkers
MeSH Terms: conditions — Muscular Atrophy, Spinal; Spinal Muscular Atrophies of Childhood

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, plasma, PBMCs, and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SMA cohort: Subjects between the ages of 2-12 years diagnosed with SMA Type I, II, or III.
- Control cohort: Healthy children between the ages of 2-12 years. These children may be either genetically-related siblings of SMA children (genetically confirmed non-carriers of SMA),or unrelated children.

SUMMARY:
The goal of this pilot study is to identify a marker or panel of markers in the blood or urine from a wide range of Spinal Muscular Atrophy (SMA) patients that segregates with measures of clinical severity. From this identification of candidate biomarkers, it is hoped that further investigations, both longitudinal natural history and clinical efficacy studies, will verify a biomarker with the sensitivity and specificity that will allow its eventual use as a validated pharmacodynamic marker or surrogate endpoint. In addition, this effort may elucidate biological pathways that may be potential therapeutic targets.

DETAILED DESCRIPTION:
Spinal Muscular Atrophy (SMA) is one of the two most common inherited children's neuromuscular disorders. There currently is no cure and no therapeutics approved to slow progression of the disease. SMA is characterized by a loss of alpha motor neurons in the spinal cord, severe atrophy of proximal muscles and progressive debility and disability due to respiratory, gastrointestinal and functional complications of the disease.

Although SMA is a relatively common orphan disease, recruitment of patients for the number of candidate therapies is expected to become rate-limiting for the development of therapeutics.

STUDY OBJECTIVES

Primary:

* To identify candidate blood and urine biochemical markers that correlate with disease severity as determined by the Modified Hammersmith Functional Motor Scale across a range of type I, type II and type III children with Spinal Muscular Atrophy (SMA) (1).

Secondary:

* To determine if there are biomarkers from types I-III SMA patients that correlate with SMA type, age at disease onset, 10-meter Timed Walk Test (ambulatory subjects only), pulmonary function, nutritional assessment, SMN protein level, SMN transcript level or SMN2 copy number.
* To determine if identified candidate biomarkers are associated with the disease state through comparison of SMA specimens with control volunteer specimens.
* To determine if there are potential biochemical pathways that may represent targets for therapeutic intervention in SMA.

ELIGIBILITY:
Inclusion Criteria:

* Age 2 to 12 years, inclusive
* In good health (other than SMA) in the judgement of the clinical investigator ar the time of assessment

Exclusion Criteria:

* Systemic or specific-organ illness
* Any known genetic condition other than SMA requiring pharmaceutical treatment
* Use of any putative SMN-enhancing medications or treatments in the past 14 days prior to enrollment
* Use of carnitine, creatine, oral albuterol or riluzole for 14 days prior to enrollment
* Use of any oral prescription medications for 14 days prior to enrollment (exceptions: anti-reflux medications, constipation or stoll softening medications, stool bulking agents, and inhaled bronchodilator medications)
* Any illness requiring treatment of antibiotics or anti-inflammatory medication within the past 14 days
* Any rash requiring treatment within the past 7 days
* Any severe asthma attack requiring treatment with oral or parenteral steroids within the past 7 days
* Any fever over 100 degrees Fahrenheit or 38 degree Celsius within the past 7 days
* Any immunization within the past 7 days
* Any injury sustained that resulted in a bone fracture or needed stitches within the past 7 days
* Any surgery within the past 7 days
* Any receipt of anesthesia within the past 7 days
* Any Emergency Room visit or hospitalization within the past 7 days
* Any stomach illness with vomiting within the past 7 days
* Any migraine headache within the past 7 days
* Participation in a clinical trial (except observational studies) within the past 7 days

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children's Hospitals Unviersity Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To identify candidate blood and urine biochemical markers that correlate with disease severity as determined by the Modified Hammersmith Functional Motor Scale across a range of type I, type II and type III children with Spinal Muscular Atrophy (SMA) | 1 year

SECONDARY OUTCOMES:
To determine if there are biomarkers from types I-III SMA patients that correlate with SMA type, age at disease onset, 10-meter Timed Walk Test, pulmonary function, nutritional assessment, SMN protein level, SMN transcript level or SMN2 copy number. | 1 year
To determine if identified candidate biomarkers are associated with the disease state through comparison of SMA specimens with control volunteer specimens. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Richard Finkel, MD, Principal Investigator — Children's Hospital of Philadelphia; Thomas Crawford, MD, Principal Investigator — Johns Hopkins University; Petra Kaufmann, MD, Principal Investigator — Columbia University
Locations (18):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Stanford, California
  - The Children's Hospital, Aurora, Colorado
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University Medical School, St Louis, Missouri
  - Columbia University SMA Clinical Research Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Medical Center - Dallas, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Canada (2):
  - Children's Hospital - London Health Sciences Center, London, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Derived] Finkel RS, Crawford TO, Swoboda KJ, Kaufmann P, Juhasz P, Li X, Guo Y, Li RH, Trachtenberg F, Forrest SJ, Kobayashi DT, Chen KS, Joyce CL, Plasterer T; Pilot Study of Biomarkers for Spinal Muscular Atrophy Trial Group. Candidate proteins, metabolites and transcripts in the Biomarkers for Spinal Muscular Atrophy (BforSMA) clinical study. PLoS One. 2012;7(4):e35462. doi: 10.1371/journal.pone.0035462. Epub 2012 Apr 27. PMID 22558154
- [Derived] Crawford TO, Paushkin SV, Kobayashi DT, Forrest SJ, Joyce CL, Finkel RS, Kaufmann P, Swoboda KJ, Tiziano D, Lomastro R, Li RH, Trachtenberg FL, Plasterer T, Chen KS; Pilot Study of Biomarkers for Spinal Muscular Atrophy Trial Group. Evaluation of SMN protein, transcript, and copy number in the biomarkers for spinal muscular atrophy (BforSMA) clinical study. PLoS One. 2012;7(4):e33572. doi: 10.1371/journal.pone.0033572. Epub 2012 Apr 27. PMID 22558076
- See also: The mission of the Spinal Muscular Atrophy Foundation is to accelerate the development of a treatment for SMA, the number one genetic killer of infants and toddlers. — http://www.smafoundation.org